CLINICAL TRIAL: NCT03262181
Title: The Acute Effects of an Isometric Loading Intervention on Lower Extremity Landing Biomechanics in Individuals With Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-1731
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Tendinopathy
Keywords: Exercise; Physical Activity; Biomechanics
MeSH Terms: conditions — Tendinopathy; Motor Activity | interventions — Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants are masked to their group assignment until the end of the study. Investigator is masked to intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Exercise Condition (Experimental): The participant will perform 5 sets of a 45-second isometric contractions at 70% of their maximum voluntary isometric contraction (MVIC). During the 45-second contraction, the participant will be provided with visual biofeedback on a computer screen (70% MVIC target line and +/- 5% error lines). The participant will be instructed to produce a level of isometric quadriceps contraction that maintains the isometric torque output line as close the target line as possible and always between the two error lines.
  Interventions: Other: Isometric Exercise
- Sham TENS Condition (Sham Comparator): Two electrodes of the Select System TENS unit (Empi, Inc., St. Paul, MN) will be placed on either side of the patellar tendon on the test limb. The same instruction script will be used for each participant, stating, "A surface electrode has been placed on either side of your patellar tendon. I will turn on the stimulation unit to emit a stimulus to your patellar tendon. This is a special sub-sensory stimulation treatment, so you will not feel anything during this period as the stimulus is set at a very low, non-detectable threshold. Please remain still during this 45-second period, letting your leg rest passively in the machine without contracting your leg muscles. After the 45-second period, the stimulation unit will be turned off and you will have a 2-minute rest period. We will repeat this same treatment/rest sequence 5 total times."
  Interventions: Other: Sham Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Isometric Exercise — 5 sets of 45-seconds quadriceps contraction, each followed by 2-minutes of rest.
  Other Names: Therapeutic Exercise
  Arms: Isometric Exercise Condition
Other: Sham Transcutaneous Electrical Nerve Stimulation — 5 sets of 45-seconds intervals without quadriceps contraction, each followed by 2-minutes of rest.
  Other Names: Sham TENS
  Arms: Sham TENS Condition

SUMMARY:
The purpose of this study is to determine differences in lower extremity landing biomechanics and real-world physical activity between individuals with patellar tendinopathy compared to individuals without patellar tendinopathy,and to determine the acute effects of an isometric loading intervention on lower extremity landing biomechanics in individuals with patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit a convenience sample of participants who meet the following overall criteria:

1. Age 15 and post-pubertal (confirmed by Pubertal Development Scale Questionnaire) - 28 years
2. Actively participating within an organized sport setting (high school, collegiate, club, competitive intramural sports) in their respective team's weekly training and competitions, quantified by a Tegner Activity Level Scale of at least 5.

Exclusion Criteria:

The following exclusion criteria will be applied to all participants:

1. Any anterior knee pain with no patellar tendon abnormality on ultrasound assessment.
2. History of any knee joint surgery ever.
3. History of other (non-knee) lower extremity surgery in the last 1 year.
4. History of lower extremity injury in last 6 months (other than patellar tendinopathy).
5. An injection (corticosteroids, plasma-rich-protein, etc.) to the patellar tendon in the last 3 months.
6. Known history of osteoarthritis or current symptoms related to osteoarthritis (i.e. stiffness, swelling).
7. Participation in formal rehabilitation for patellar tendinopathy in prior 3 months
8. Known neurological disorders, including: stroke, multiple sclerosis, ALS, diabetic neuropathy, epilepsy, traumatic brain injury resulting in loss of consciousness, concussion within the last 6 months, cranial neural surgery, balance disorders.
9. Use of pacemaker or another implantable electronic device.
10. History of cardiac arrhythmia or any cardiac condition.
11. History of psychiatric disorder. *
12. History of cancer in the brain or thigh musculature.
13. Pubertal Development Scale Score < 12 (Stages 1-4)

    * Note: Rationale for exclusion of individuals with a history of psychiatric disorders is that these individuals may have taken or be taking pharmacological agents that could affect pain or neuromuscular control.

Ages: 15 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Difference in the change in mean internal knee extension moment during landing between groups | Pre- and post-intervention condition (~30 minutes)
  Angular force or moment will be measured in Nm/kg*m where "Nm" represents angular force and "kg*m" represents normalization to body weight and height.
Difference in the change in mean internal hip flexion moment during landing between groups | Pre- and post-intervention condition (~30 minutes)
  Angular force or moment will be measured in Nm/kg*m where "Nm" represents angular force and "kg*m" represents normalization to body weight and height.
Difference in the change in mean peak vertical ground reaction force during landing between groups | Pre- and post-intervention condition (~30 minutes)
  Vertical ground reaction force will be measured in N(BW) where "N" is a measure of force and "BW" represents normalization to body weight.
Difference in the change in mean peak vertical ground reaction force loading rate during landing between groups | Pre- and post-intervention condition (~30 minutes)
  Vertical ground reaction force loading rate will be measured in N(BW)/s where "N" is a measure of force and "BW" represents normalization to body weight and "s" is the time unit seconds.
Difference in the change in mean peak patellar tendon force during landing between groups | Pre- and post-intervention condition (~30 minutes)
  Patellar tendon force will be measured in N(BW) where "N" is a measure of force and "BW" represents normalization to body weight.

SECONDARY OUTCOMES:
Difference in average steps-per-day between groups | Day 1 - Day 7
  Steps-per-day calculated by an ActiGraph GT9X Link Accelerometer (ActiGraph Corporation, Pensacola, FL) wearable physical activity device worn at the hip using a belt clip.
Difference in average minutes of moderate-to-vigorous physical activity (MVPA) between groups | Day 1 - Day 7
  MVPA calculated by an ActiGraph GT9X Link Accelerometer (ActiGraph Corporation, Pensacola, FL) wearable physical activity device worn at the hip using a belt clip.
Difference in change in anterior knee pain (self-reported via visual analog scale (0-10)) between groups | Pre- and post-intervention condition (~10 minutes)
  A standard visual analog scale (0-10) will be utilized to assess pain, where 0=complete absence of pain and 10=worst pain imaginable (higher scores indicate worse pain). This scale will be delivered verbally and the participants will respond verbally.

CONTACTS AND LOCATIONS:
Overall Officials: Darin A Padua, PhD, ATC, Study Chair — Professor and Department Chair; Laura E Stanley, DPT, Principal Investigator — Graduate Research Assistant
Locations (1):
- Sports Medicine Research Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided